CLINICAL TRIAL: NCT00551070
Title: A Phase II Trial of AZD6244 (NSC# 748727) in Women With Recurrent Low-Grade Serous Carcinoma of the Ovary or Peritoneum
Brief Title: Selumetinib Sulfate in Treating Woman With Recurrent Low-Grade Ovarian Cancer or Peritoneum Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00604; NCI-2009-00604 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000563965; GOG-0239 (Other: NRG Oncology); GOG-0239 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2007-10-22; First posted 2007-10-30 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Borderline Ovarian Serous Tumor; Low Grade Ovarian Serous Adenocarcinoma; Micropapillary Serous Carcinoma; Primary Peritoneal Carcinoma; Primary Peritoneal Low Grade Serous Adenocarcinoma; Recurrent Borderline Ovarian Surface Epithelial-Stromal Tumor
MeSH Terms: conditions — Cystadenocarcinoma, Serous | interventions — AZD 6244

ARMS (1):
- Treatment (selumetinib sulfate) (Experimental): Patients receive selumetinib sulfate PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Selumetinib; Drug: Selumetinib Sulfate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate

SUMMARY:
This phase II trial studies the side effects and how well selumetinib sulfate works in treating patients with low-grade ovarian cancer that has come back (recurrent). Selumetinib sulfate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the tumor response rate of patients on AZD6244 (selumetinib sulfate) (NSC #748727).

II. To examine the acute toxicity of AZD6244 (NSC #748727) during the first course of treatment using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

III. To define the pharmacokinetic profile for AZD6244, 100 mg administered orally twice daily.

SECONDARY OBJECTIVES:

I. To examine the toxicity of AZD6244 (NSC #748727) using the 21 major categories of the CTCAE version 3.0.

II. To examine the dose and number of courses of AZD6244 (NSC #748727) given. III. To estimate the progression free survival, and overall survival of women receiving AZD6244 (NSC #748727).

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To examine deoxyribonucleic acid (DNA) isolation with sequencing of braf, and ras mutation analysis and to explore their relationship with tumor response with AZD6244 (NSC #748727).

II. To examine protein levels of phosphorylated (p)-ERK/ERKERK) and explore their relationship with tumor response in patients treated with AZD6244 (NSC #748727).

OUTLINE:

Patients receive selumetinib sulfate orally (PO) twice a day (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for correlative and pharmacokinetic studies and to analyze selumetinib sulfate peak concentrations and the corresponding peak time values. Previously collected archived tumor tissue samples are obtained to determine protein levels of p-ERK/ERKERK, DNA isolation and sequencing of BRAF and ras mutation analysis by immunohistochemistry (IHC).

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then once a year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than 18 with the following tumors are included in the study:

  * Patients initially diagnosed with low-grade serous ovarian or peritoneal carcinoma that recur as low grade serous carcinoma (invasive micropapillary serous carcinoma or invasive grade I serous carcinomas as defined by Gynecologic Oncology Group [GOG], International Federation of Gynecology and Obstetrics [FIGO] World Health Organization [WHO] or Silverberg)
  * Patients initially diagnosed with serous borderline ovarian or peritoneal carcinoma that recur as low grade serous carcinoma (invasive micropapillary serous carcinoma or invasive grade I serous carcinomas as defined by GOG, FIGO WHO or Silverberg)
* Patients must have measurable disease:

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each "target" lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Patient must have documented low grade serous carcinoma (invasive micropapillary serous); confirmation must occur before patient is considered eligible for the trial

  * Patients whose primary tumor was low-grade serous ovarian or peritoneal carcinoma must have a pretreatment sample of their tumor from their primary or recurrent tumor that documents low grade serous carcinoma (invasive micropapillary serous)
  * Patients whose primary tumor was serous borderline ovarian or peritoneal carcinoma must have a pretreatment sample of their tumor from their recurrent tumor that documents low grade serous carcinoma (invasive micropapillary serous)
* Creatinine CTCAE grade 0-1 (< 1.5 x upper limit of normal [ULN])
* Bilirubin CTCAE grade 0-1 (< 1.5 x ULN)
* Transaminases CTCAE grade 0-1 (< 2.5 x ULN)
* Neutrophil CTCAE grade 0-1 (>= 1500/mcl)
* Platelets CTCAE grade 0-1 (>= 100,000/mcl)
* Neuropathy =< CTCAE grade 1
* No restrictions on prior therapy; patients cannot have previously received AZD6244
* Patients of childbearing potential must have a negative pregnancy test and must agree to practice an effective means of birth control prior to study entry, for the duration of study participation, and for four weeks after dosing with AZD6244 ceases
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have a GOG performance status of 0 or 1

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or its excipient Captisol
* Previous mitogen-activated protein kinase (MEK) inhibitor use
* Patients with corrected QT (QTc) interval > 450 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class III and IV definitions are excluded
* Required use of a concomitant medication that can prolong the QT interval
* Patients should not receive any drugs known to affect or with the potential to affect selected CYP450 isoenzymes
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of AZD6244 on the developing human fetus at the recommended therapeutic dose are unknown; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with AZD6244
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2013-07-23 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Farley, Principal Investigator — NRG Oncology
Locations (49):
- United States (49):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Farley J, Brady WE, Vathipadiekal V, Lankes HA, Coleman R, Morgan MA, Mannel R, Yamada SD, Mutch D, Rodgers WH, Birrer M, Gershenson DM. Selumetinib in women with recurrent low-grade serous carcinoma of the ovary or peritoneum: an open-label, single-arm, phase 2 study. Lancet Oncol. 2013 Feb;14(2):134-40. doi: 10.1016/S1470-2045(12)70572-7. Epub 2012 Dec 21. PMID 23261356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/22/2008 and closed to accrual on 1/31/2011 (suspended from 1/4/2010 to 8/9/2010).
Groups:
- AZD6244: AZD6244 (NSC #748727) 100 mg orally BID until disease progression or adverse effects prohibit further therapy (1 cycle =28 days)
Period: Overall Study
Arm/Group | AZD6244
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | AZD6244
Number analyzed (Participants) | 52
Age, Customized [Number; unit: participants]
  20-29 years | 3
  30-39 years | 11
  40-49 years | 8
  50-59 years | 17
  60-69 years | 9
  70-79 years | 4
  80-89 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by (Response Evaluation Criteria in Solid Tumors) RECIST 1.0
Time Frame: Every other cycle
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | AZD6244
Number analyzed (Participants) | 52
percentage of patients | 15.4 [7.9 to 26.1]

2. Secondary Outcome: Progression-free Survival
Time Frame: Every other cycle
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD6244
Number analyzed (Participants) | 52
months | 11.3 [6.2 to 12.9]

3. Secondary Outcome: Number of Courses Received
Time Frame: Every cycle
Population: Eligible and Treated Patients. Two patients still on study and have received 68 and 79 cycles of treatment.
Measure: Median (Inter-Quartile Range); unit: courses
Arm/Group | AZD6244
Number analyzed (Participants) | 52
courses | 5 [2 to 14]

4. Primary Outcome: Adverse Events (Grade 3 or Higher) During First Cycle of Treatment
Time Frame: Cycle 1
Population: Eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AZD6244
Number analyzed (Participants) | 52
percentage of patients
  Leukopenia | 0 [0 to 7]
  Thrombocytopenia | 0 [0 to 7]
  Neutropenia | 0 [0 to 7]
  Anemia | 2 [0 to 10]
  Allergy/Immunology | 0 [0 to 7]
  Auditory/Ear | 0 [0 to 7]
  Cardiac | 2 [0 to 10]
  Coagulation | 0 [0 to 7]
  Constitutional | 4 [0 to 13]
  Dermatologic | 12 [4 to 23]
  Gastrointestinal | 13 [6 to 26]
  Genitourinary/Renal | 2 [0 to 10]
  Hemorrhage | 0 [0 to 7]
  Infection | 0 [0 to 7]
  Lymphatics | 0 [0 to 7]
  Metabolic | 0 [0 to 7]
  Musculoskeletal | 0 [0 to 7]
  Neurosensory | 0 [0 to 7]
  Other Neurological | 0 [0 to 7]
  Ocular/Visual | 0 [0 to 7]
  Pain | 4 [0 to 13]
  Pulmonary | 4 [0 to 13]

5. Primary Outcome: Area Under the Curve (AUC) for AZD6244, 100 mg Administered Orally Twice Daily.
Time Frame: Pre-dose, and 1, 3, and 6 hours after administration of drug on Day 7 after the start of AZD6244 treatment
Population: Eligible and Treated Patients with all pharmacokinetic time points available
Measure: Median (Inter-Quartile Range); unit: ng x hr/mL
Arm/Group | AZD6244
Number analyzed (Participants) | 41
ng x hr/mL | 2419 [1673 to 3186]

6. Primary Outcome: Maximum Concentration (Cmax) for AZD6244, 100 mg Administered Orally Twice Daily.
Time Frame: Pre-dose, and 1, 3, and 6 hours after administration of drug on Day 7 after the start of AZD6244 treatment
Population: Eligible and Treated Patients with at least one post-dose pharmacokinetic time point available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | AZD6244
Number analyzed (Participants) | 42
ng/mL | 585 [371 to 1100]

7. Secondary Outcome: Overall Survival
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD6244
Number analyzed (Participants) | 52
Months | 32.4 [17.7 to 39.3]

ADVERSE EVENTS:
Time Frame: Study Treatment
Description: Includes all adverse events reported (grade 1-5) regardless of attribution.
Arm/Group | AZD6244
Serious Adverse Events (participants affected / at risk) | 33/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6244 (N=52)
Leukocytes (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Prolonged Qtc Interval (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 1
Weight Gain (General disorders) | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 2
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 4
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Stricture, Gi - Biliary Tree (Gastrointestinal disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2
Inf Unknown Anc: Wound (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 1
Alt (Metabolism and nutrition disorders) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 1
Pain: Back (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 4
Ards (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6244 (N=52)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Rhinitis (Immune system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 4
Neutrophils (Blood and lymphatic system disorders) | 10
Platelets (Blood and lymphatic system disorders) | 6
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 11
Hemoglobin (Blood and lymphatic system disorders) | 28
Prolonged Qtc Interval (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 5
Inr (Vascular disorders) | 2
Constitutional Symptoms - Other (General disorders) | 2
Sweating (General disorders) | 1
Weight Gain (General disorders) | 11
Fever (General disorders) | 5
Weight Loss (General disorders) | 2
Rigors/Chills (General disorders) | 3
Fatigue (General disorders) | 39
Insomnia (General disorders) | 6
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 10
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 31
Dry Skin (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 2
Hand-Foot (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 1
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Distention (Gastrointestinal disorders) | 4
Taste Alteration (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 4
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 9
Mucositis (Clinical Exam) - Esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 25
Anorexia (Gastrointestinal disorders) | 12
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 35
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 41
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 3
Hemorrhage, Gu - Vagina (Vascular disorders) | 2
Hemorrhage/Pulmonary - Bronchopulmonary Nos (Vascular disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 2
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 4
Hemorrhage, Gi - Colon (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 2
Infection - Other (Infections and infestations) | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 1
Inf Unknown Anc: Pharynx (Infections and infestations) | 1
Inf Unknown Anc: Bronchus (Infections and infestations) | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Lymphocele (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 24
Edema: Head And Neck (Blood and lymphatic system disorders) | 4
Ast (Metabolism and nutrition disorders) | 24
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 5
Proteinuria (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Ggt (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 20
Alkaline Phosphatase (Metabolism and nutrition disorders) | 16
Bilirubin (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 18
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 5
Mood Alteration - Anxiety (Nervous system disorders) | 9
Tremor (Nervous system disorders) | 1
Speech Impairment (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Neuropathy-Sensory (Nervous system disorders) | 20
Ocular/Visual - Other (Eye disorders) | 2
Watery Eye (Eye disorders) | 1
Dry Eye (Eye disorders) | 2
Blurred Vision (Eye disorders) | 4
Pain - Other (General disorders) | 2
Pain: Urethra (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 3
Pain: Head/Headache (General disorders) | 9
Pain: Neck (General disorders) | 1
Pain: Intestine (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 8
Pain: Back (General disorders) | 7
Pain: Joint (General disorders) | 5
Pain: Bladder (General disorders) | 1
Pain: Pain Nos (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 20
Pain: Skin (General disorders) | 1
Pain: Cardiac/ Heart (General disorders) | 1
Pain: Muscle (General disorders) | 5
Pain: Anus (General disorders) | 1
Pain: Sinus (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Study began with 100mg BID mix & drink (MD) formulation. AstraZeneca (AZ) switched to hydrogen-sulfate capsule (HC). AZ deemed 100mg BID MD equivalent to 50mg BID HC. As of 12/31/2010, patients got 50mg BID HC; four patients were on treatment then.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less